CLINICAL TRIAL: NCT06807281
Title: A Phase 3, Multicenter, Long-Term, Open Label Study Evaluating the Safety and Efficacy of Abrocitinib, With or Without Topical Medications Administered to Pediatric Participants Aged 2 Years and Older With Moderate-to-Severe Atopic Dermatitis
Brief Title: A Long-term Study of the Medicine Called Abrocitinib in Children Aged 2 Years and Older With Moderate to Severe Eczema
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: B7451031; 2023-509124-18-00 (Registry Identifier: CTIS (EU))
Record Dates: First submitted 2025-01-29; First posted 2025-02-04 (Actual); Last update posted 2026-01-09 (Actual); Status verified 2026-01

CONDITIONS: Atopic Dermatitis
Keywords: eczema; atopic dermatitis
MeSH Terms: conditions — Dermatitis, Atopic; Eczema | interventions — abrocitinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Extension (Experimental): Patients who have completed other abrocitinib studies
  Interventions: Drug: Abrocitinib
- De novo (Experimental): Patients who have not participated other abrocitinib studies
  Interventions: Drug: Abrocitinib

INTERVENTIONS:
Drug: Abrocitinib — Abrocitinib administered as liquid oral suspension.
  Other Names: PF-04965842

SUMMARY:
This 24-month study will assess the long-term safety and efficacy of liquid abrocitinib oral suspension with or without topical medications in children 2 years of age or older with moderate-to-severe atopic dermatitis. The study will enroll two groups: participants who have completed other abrocitinib studies and participants who have never participated in abrocitinib studies.

DETAILED DESCRIPTION:
Phase 3, open-label study to assess the long-term safety and efficacy of liquid abrocitinib oral suspension with or without topical medications in children ≥2 years of age with moderate-to-severe atopic dermatitis (AD). This study will enroll participants in two cohorts: an extension cohort of participants who previously completed prior abrocitinib studies, and a de novo cohort of participants (6 to <12 years of age) who have not participated in previous abrocitinib studies. Study duration will be up to 2 years (or commercial availability, whichever occurs earlier). The study will enroll a maximum of approximately 500 participants with moderate-to-severe Atopic Dermatitis from study sites globally (extension cohort will enroll up to 320 participants; de novo cohort will enroll approximately 180 participants). All participants will receive the study intervention abrocitinib oral suspension.

ELIGIBILITY:
Inclusion Criteria for the Extension Cohort:

1. Participants who have completed the treatment phase of the qualifying parent study (age 2 to <12 years old).

• No contraception methods are required for male participants. Female participants must not be pregnant or breastfeeding and, if the participant is of child-bearing potential, must use a highly effective form of contraception (i.e., abstinence) during the study intervention period and for at least 28 days after the last dose of study intervention.

Inclusion Criteria for the De Novo Cohort:

Age

1. Children aged 6 to <12 years at the time of informed consent/assent.

   • No contraception methods are required for male participants.

   Disease Characteristics:
2. Participants who meet all of the following AD criteria:

   * A documented diagnosis of chronic AD for at least 6 months prior to screening and confirmed at screening and baseline visits according to the Hanifin and Rajka criteria; and
   * A diagnosis of moderate-to-severe AD at the baseline visit (must fulfill all of the following criteria: BSA ≥10%, vIGA ≥3, EASI ≥16, and WI-NRS ≥4); and
   * Documented history (within 6 months of the screening visit) of inadequate response to treatment with topical medical therapy for AD (eg, TCS and TCI), for at least 4 weeks and are candidates for systemic therapy.

   Other Inclusion Criteria:
3. Body weight ≥15 kg

Exclusion Criteria for the Extension Cohort:

Medical Conditions:

1. Any medical or psychiatric condition including any active suicidal ideation in the past year or suicidal behavior in the past 5 years or laboratory abnormality that may increase the risk of study participation or, in the investigator's judgment, make the participant inappropriate for the study.

   If the participant has SDQ total score ≥17, the investigator should exclude the child or refer them to a pediatric MHP to determine if it is safe to participate in the study. A copy or summary of the evaluation should be placed in the site source documents.

   Prior/Concomitant Therapy:
2. Required use of any prohibited concomitant treatments outlined in Section 6.9.3 and Appendix 9 of study protocol.
3. Required vaccination with live attenuated vaccines during study treatment and for 6 weeks after discontinuing study treatment.

   Diagnostic Assessments:
4. Ongoing adverse event in the parent studies which in the opinion of the investigator, or sponsor, is an ongoing safety concern OR the participant is currently triggering safety monitoring criteria.
5. Discontinued from treatment early in the parent studies OR triggered a discontinuation criterion at any point during the parent studies OR meets exclusion criteria from the parent studies which in the opinion of the investigator, or sponsor, is an ongoing safety concern.

Exclusion Criteria for the De Novo Cohort

Medical Conditions:

1. Any medical or psychiatric condition including any active suicidal ideation in the past year or suicidal behavior in the past 5 years or laboratory abnormality that may increase the risk of study participation or, in the investigator's judgment, make the participant inappropriate for the study.

   If the participant has SDQ total score ≥17, the investigator should exclude them or refer the child to a pediatric MHP to determine if it is safe to participate in the study. A copy or summary of the evaluation should be placed in the site source documents.
2. Have any of the following medical conditions:

   * Infections:

     * Skin infections that require treatment with systemic antimicrobials within 2 weeks prior to Day 1 (baseline) or have superficial skin infections within 1 week of Day 1.
     * History of systemic infection requiring hospitalization or parenteral antimicrobial therapy or as otherwise judged clinically significant by the investigator within 1 month prior to Day 1.
     * Have a history (single episode) of disseminated herpes zoster or disseminated herpes simplex, or a recurrent localized, dermatomal herpes zoster.
     * Infection with HIV, hepatitis B, and/or hepatitis C
     * Evidence of active TB or inadequately treated latent TB.
   * Skin Conditions:

     - Including but not limited to psoriasis, seborrheic dermatitis or lupus on Day 1 that would interfere with evaluation of AD or response to treatment.
   * Other Conditions:

     * Documented history of skeletal dysplasia.
     * Documented history of retinal detachment.
     * History of or conditions associated with thrombocytopenia, coagulopathy or platelet dysfunction.
     * Prior history of leukemia, lymphoma, sarcoma or any other malignancy.
     * Immunodeficiency disorder or a first-degree relative with a hereditary immunodeficiency.
     * Any other medical conditions that in the investigator's judgment make the participant inappropriate for the study.

   Prior/Concomitant Therapy:
3. Prior treatment with a systemic JAK inhibitor for AD.
4. Live attenuated vaccination within 6 weeks prior to Day 1 or require vaccination with live attenuated vaccines during treatment or within 6 weeks after the last dose of study intervention.
5. Concomitant use of strong inhibitors and inducers of CYP2C19 enzymes and strong inducers of CYP2C9 enzymes is not allowed in the study.

   Prior/Concurrent Clinical Study Experience:
6. Previous administration of an investigational drug within 30 days or 5 half lives, whichever is longer, of Day 1.

   Diagnostic Assessments:
7. Hepatic and/or renal and/or hematological abnormalities defined as:

   * AST >2 x ULN
   * Hemoglobin <10 g/dL
   * ALT >2 x ULN
   * ANC <1000/mm3
   * Total bilirubin ≥1.5 x ULN
   * ALC <500/mm3
   * eGFR <60 mL/min/1.73 m2
   * Platelets <150,000 /mm3

   Other Exclusion Criteria:
8. Investigator site staff directly involved in the conduct of the study and their family members, site staff otherwise supervised by the investigator, and sponsor and sponsor delegate employees directly involved in the conduct of the study and their family members.

Ages: 2 Years to 11 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 500 (Estimated)
Dates: Start 2025-12-02 (Actual); Primary Completion 2032-02-22 (Estimated); Study Completion 2032-02-22 (Estimated)

PRIMARY OUTCOMES:
Number of Participants with Treatment-Emergent Adverse Events (TEAEs), Serious Adverse Events (SAEs), and adverse events (AEs) that lead to study discontinuation | 0-24 months
  The number of the treatment emergent adverse events, serious adverse events and adverse events leading to discontinuation among patients with moderate-to-severe disease treated with abrocitinib regardless of discontinuation from study treatment.

SECONDARY OUTCOMES:
Number of Participants With Clinically Significant Laboratory Abnormalities | 0-24 months
  The number of clinically significant laboratory abnormalities among participants with moderate-to-severe disease treated with abrocitinib.
Response based on achieving Validated Investigator's Global Assessment (vIGA) score of clear (0) or almost clear (1) (on a 5-point scale) and a 2 -point reduction from baseline at all scheduled time points | Baseline, 24 months
  Proportion of responders based on vIGA at all scheduled time points in patients with moderate-to-severe disease treated with abrocitinib
Percentage of Response based on achieving a ≥4 point improvement from baseline in the Worst Itch Numerical Rating Scale (WI-NRS) at all scheduled time points in participants aged ≥2 to <6 years | 0-24 months
  Percentage of responders based on achieving an improvement ≥4 points from baseline at all scheduled time points in the WI-NRS (in patients aged ≥2 to <6 years) with moderate-to-severe disease treated with abrocitinib.
Percentage of Response based on achieving a ≥4-point improvement from baseline in the WSI-NRS at all scheduled time points in participants aged ≥6 to 12 years | 0-24 months
  Percentage of responders based on achieving an improvement ≥4 points from baseline at all scheduled time points in the WSI-NRS (in patients aged ≥6 to 12 years) with moderate-to-severe disease treated with abrocitinib.
Percentage of Responders based on achieving Eczema Area and Severity Index (EASI)-50, EASI-90 and EASI-100 at all scheduled time points in participants with moderate-to-severe disease treated with abrocitinib | 0-24 months
  Percentage of response based on achieving ≥50%, ≥90%, 100% improvement from parent study baseline in the EASI total score (EASI-50, EASI-90, EASI-100) at all scheduled time points.
Percent Change from Baseline (CFB) in EASI total score at all scheduled time points. | 0-24 months
  Mean percent CFB in EASI total score at all scheduled time points in patients with moderate-to-severe disease treated with abrocitinib
Percentage of Participants with Flares | 0-24 months
  Percentage of participants reporting flares in patients with moderate-to-severe disease treated with abrocitinib.
CFB in the percentage Body Surface Area (BSA) affected at all scheduled time points | 0-24 months
  Mean CFB in BSA affected at all scheduled time points in patients with moderate-to-severe disease treated with abrocitinib.
CFB in Children's Dermatology Life Quality Index (CDLQI) at all scheduled time points. | 0-24 months
  Mean CFB in CDLQI at all scheduled time points in participants aged ≥4 to <16 years with moderate-to-severe disease treated with abrocitinib.
CFB in in Infants' Dermatitis Quality of Life (IDQOL) Index at all scheduled time points | 0-24 months
  Mean CFB in IDQOL Index or CDQLI depending on age at all scheduled time points in participants aged <4 years with moderate-to-severe disease treated with abrocitinib
CFB in Patient-Oriented Eczema Measure (POEM) at all scheduled time points | 0-24 months
  Mean CFB in POEM at all scheduled time points in participants with moderate-to-severe disease treated with abrocitinib.
CFB in Dermatitis Family Impact (DFI) at all scheduled time points | 0-24 months
  Mean CFB in DFI at all scheduled time points in participants with moderate-to-severe disease treated with abrocitinib.
CFB in Patient Global Impression of Severity (PGIS) at all scheduled time points | 0-24 months
  Mean CFB in PGIS (in patients aged 6 to <12 years) at all scheduled time points in patients with moderate-to-severe disease treated with abrocitinib.
CFB in Observer Reported Global Impression of Severity (OGIS) at all scheduled time points | 0-24 months
  Mean CFB in OGIS (in patients aged 2 to <6 years) at all scheduled time points in patients with moderate-to-severe disease treated with abrocitinib
CFB in the the EuroQol- 5 Dimension Youth (EQ-5D-Y) | 0-24 months
  Mean CFB in EQ-5D-Y at all scheduled time points in patients with moderate-tosevere AD treated with abrocitinib versus placebo.
Number of topical corticosteroid and /or topical calcineurin inhibitor free days | 0-24 months
  Mean number of days free from topical corticosteroids and /or topical calcineurin inhibitor use in patients with moderate-to-severe disease treated with abrocitinib.
Percentage of Participants Achieving satisfactory response in Tdap/DTaP and/or pneumococcal antibody titers as appropriate in participants who receive Tdap/DTaP and/or pneumococcal vaccinations | 0-24 months
  For patients that receive Tdap/ DTap and/or pneumococcal vaccinations during the study, the proportion of patients treated with abrocitinib who achieve satisfactory immunogenicity at 4 weeks after receiving the vaccinations.

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (18):
- United States (6):
  - Cahaba Dermatology & Skin Health Center, Birmingham, Alabama
  - Arkansas Research Trials, North Little Rock, Arkansas
  - Solutions Through Advanced Research, Jacksonville, Florida
  - Miami Dermatology and Laser Research, Miami, Florida
  - Dawes Fretzin Clinical Research Group, LLC, Indianapolis, Indiana
  - Tribe Clinical Research, LLC, Greenville, South Carolina
- Universitätsklinikum Münster, Münster, North Rhine-Westphalia, Germany
- Hungary (2):
  - Pécsi Tudományegyetem Klinikai Központ, Pécs, Baranya
  - Clinexpert Kft., Budapest, Pest County
- Japan (4):
  - Queen's square Medical Facilities Queen's square Dermatology and Allergology, Yokohama, Kanagawa
  - Dermatology and Ophthalmology Kume Clinic, Sakai, Osaka
  - Sasamoto Children's Clinic, Setagaya-ku, Tokyo
  - Fukuoka National Hospital, Fukuoka
- Poland (2):
  - Centrum Medyczne Evimed, Warsaw, Masovian Voivodeship
  - Dermedic Jacek Zdybski, Ostrowiec Świętokrzyski, Świętokrzyskie Voivodeship
- Spain (3):
  - CHUS - Hospital Clinico Universitario, Santiago de Compostela, A Coruña [LA Coruña]
  - Hospital General de Granollers, Granollers, Barcelona
  - Hospital Universitario Miguel Servet, Zaragoza

IPD SHARING:
Plan to Share IPD: Yes
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.
URL: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=B7451031